CLINICAL TRIAL: NCT01010971
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Clinical Trial to Assess the Efficacy and Safety of Ciclesonide HFA Nasal Aerosol (160 μg Once Daily and 80 μg Once Daily) for the Treatment of Seasonal Allergic Rhinitis (SAR) to Mountain Cedar in Subjects 12 Years and Older
Brief Title: Clinical Trial to Assess the Efficacy and Safety of Ciclesonide Hydrofluoroalkane (HFA) Nasal Aerosol for the Treatment of Seasonal Allergic Rhinitis (SAR) to Mountain Cedar in Subjects 12 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-634
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Mountain Cedar
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ciclesonide HFA Nasal Aerosol 160 μg (Experimental): 160 μg once daily
  Interventions: Drug: Ciclesonide HFA 160 μg
- Ciclesonide HFA Nasal Aerosol 80 μg (Experimental): 80 μg once daily
  Interventions: Drug: Ciclesonide HFA 80 μg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide HFA 160 μg — Ciclesonide HFA Nasal Aerosol 160 μg once daily
  Arms: Ciclesonide HFA Nasal Aerosol 160 μg
Drug: Ciclesonide HFA 80 μg — Ciclesonide HFA Nasal Aerosol 80 μg once daily
  Arms: Ciclesonide HFA Nasal Aerosol 80 μg
Drug: Placebo — Placebo HFA Nasal Aerosol once daily
  Arms: Placebo

SUMMARY:
This clinical research study will evaluate the safety and effectiveness of two doses of an investigational medication (ciclesonide nasal aerosol) for the treatment of subjects with of seasonal allergic rhinitis (SAR). The study will consist of a Screening Period to confirm study eligibility, followed by a Single-Blind Placebo Run-in period to acclimate subjects to the proper use of the study medication and to assess the subject's severity of SAR symptoms, followed by a 2-week double-blind treatment period to assess the safety and effectiveness of the study medication when given to eligible subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. This study will consist of a Screening Period, followed by a Single-Blind Placebo Run-in period. The Double-blind Treatment period (14±2 days) will begin at randomization/Day 1 and consist of an interim visit 7±1 days after randomization, and an End of Study (EOS)/Early Termination (ET) visit. All subjects will have either a telephone contact, or in some cases an in-clinic visit, 7±2 days after their last study visit. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, medical history, and clinical laboratory values (Hematology, Chemistries and Urinalysis). If any of the Hematology, Chemistries, or Urinalysis are not within the clinical laboratory's reference range, then the subject can be included only if the Investigator judges the deviations to be not clinically significant.
* A history of SAR to Mountain Cedar for a minimum of two years immediately preceding the study Screening Visit. The SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and in the Investigator's judgment (through exposure to allergen) is expected to require treatment throughout the entire study period.
* A demonstrated sensitivity to Mountain Cedar known to induce SAR through a standard skin prick test administered at screening. A positive test is defined as a wheal diameter at least 5 mm larger than the control wheal (normal saline) for the skin prick test.
* Subject, if female 65 years of age or younger, must have a negative serum pregnancy test. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study and will continue its use throughout the study and for thirty days following study participation; Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study; Abstinence.
* Subject or parent/guardian must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator as well as accurately complete both the AR diary and RQLQ(S).

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; nasal ulcers or perforations; or surgery and atrophic rhinitis or rhinitis medicamentosa (all within the last 60 days prior to the Screening Visit).
* Participation in any investigational drug trial within the 30 days preceding the Screening Visit or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, chronic sinusitis, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit .
* History of alcohol or drug abuse within two years preceding the Screening Visit.
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Plans to travel outside the study area (the known pollen area for the investigative site) for more than 24 hours during the Run-in period.
* Plans to travel outside the study area (the known pollen area for the investigative site) for 2 or more consecutive days between Randomization Visit and the final Treatment Visit.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drugs (eg, theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists is acceptable.
* Use of any disallowed concomitant medications within the prescribed (per protocol) time period prior to the Screening Visit and expected use during treatment period.
* Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit. Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit and is expected to continue throughout the trial.
* Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Previous participation in an intranasal ciclesonide HFA nasal aerosol study.
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit.
* Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Study participation by clinical investigator site employees and/or their immediate relatives.
* Study participation by more than one subject from the same household at the same time.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial:

  * impaired hepatic function including alcohol-related liver disease or cirrhosis;
  * history of ocular disturbances eg, glaucoma or posterior subcapsular cataracts;
  * any systemic infection;
  * hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism);
  * gastrointestinal disease;
  * malignancy (excluding basal cell carcinoma);
  * current neuropsychological condition with or without drug therapy.
* Any condition that, in the judgement of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Allergy and Asthma Associates, Austin, Texas
  - Sinus Clinical Research LLC, Austin, Texas
  - Central Texas Health Research Corporation, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Southwest Allergy and Asthma Research Center, Pa, San Antonio, Texas
  - Sylvana Research, San Antonio, Texas
  - San Antonio, Texas

REFERENCES:
- [Result] Ratner PH, Andrews C, Martin B, Howland W, Desai SY, Huang H, Hinkle J, Bode F. A study of the efficacy and safety of ciclesonide hydrofluoroalkane nasal aerosol in patients with seasonal allergic rhinitis from mountain cedar pollen. Allergy Asthma Proc. 2012 Jan-Feb;33(1):27-35. doi: 10.2500/aap.2012.33.3490. PMID 22370531

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo once daily
Period: Overall Study
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Started | 225 | 226 | 220
Completed | 222 | 218 | 207
Not Completed | 3 | 8 | 13
Not completed — Adverse Event | 2 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 5
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Other | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo | Total
Number analyzed (Participants) | 225 | 226 | 220 | 671
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 21 | 10 | 51
  Between 18 and 65 years | 198 | 194 | 202 | 594
  >=65 years | 7 | 11 | 8 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (14.4) | 39.8 (14.7) | 41.0 (13.5) | 40.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 140 | 129 | 398
  Male | 96 | 86 | 91 | 273
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 (43.6) | 89 (39.4) | 100 (45.5) | 287 (42.8)
  Not Hispanic or Latino | 127 (56.4) | 137 (60.6) | 120 (54.5) | 384 (57.2)
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 207 | 191 | 191 | 589
  Black/African American | 13 | 26 | 23 | 62
  Asian | 3 | 7 | 5 | 15
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiin or Other Pacific Islander | 1 | 1 | 0 | 2
  Multiple | 0 | 1 | 0 | 1
  Other | 1 | 0 | 0 | 1
Baseline Reflective Total Nasal Symptom Score (rTNSS) [Mean (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 9.33 (1.78) | 9.47 (1.80) | 9.34 (1.76) | 9.38 (1.78)
    PM | 9.20 (1.97) | 9.21 (2.11) | 9.21 (1.92) | 9.21 (2.00)
    AM and PM | 9.26 (1.80) | 9.34 (1.88) | 9.28 (1.77) | 9.29 (1.82)
Baseline Instantaneous Total Nasal Symptom Score (iTNSS) [Mean (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 8.77 (2.10) | 8.73 (2.18) | 8.69 (2.19) | 8.73 (2.15)
    PM | 8.51 (2.29) | 8.49 (2.35) | 8.36 (2.38) | 8.45 (2.34)
    AM and PM | 8.64 (2.14) | 8.60 (2.15) | 8.53 (2.21) | 8.59 (2.16)
Baseline Baseline Reflective Ocular Symptom Score (rTOSS) in Subjects with rTOSS ≥5.0 [Mean (Standard Deviation); unit: units on a scale] — TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TOSS symptom scores assess symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 7.09 (1.24) | 7.17 (1.24) | 6.99 (1.21) | 7.09 (1.23)
    PM | 7.00 (1.30) | 7.10 (1.25) | 6.94 (1.30) | 7.01 (1.28)
    AM and PM | 7.04 (1.22) | 7.13 (1.19) | 6.97 (1.19) | 7.05 (1.20)
Baseline Instantaneous Total Ocular Symtom Score (iTOSS) in Subjects with iTOSS ≥5.0 [Mean (Standard Deviation); unit: units on a scale] — TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale
    AM | 7.07 (1.20) | 7.07 (1.26) | 7.05 (1.14) | 7.06 (1.20)
    PM | 6.90 (1.35) | 6.88 (1.39) | 6.92 (1.20) | 6.90 (1.31)
    AM and PM | 6.99 (1.21) | 6.97 (1.24) | 6.99 (1.07) | 6.98 (1.17)
Baseline Reflective Nasal Symptom Score (rNSS) [Mean (Standard Deviation); unit: unit on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  unit on a scale
    AM sneezing | 2.04 (0.71) | 2.10 (0.74) | 2.06 (0.70) | 2.07 (0.72)
    AM runny nose | 2.43 (0.54) | 2.43 (0.57) | 2.42 (0.55) | 2.43 (0.55)
    AM nasal itching | 2.29 (0.59) | 2.38 (0.54) | 2.31 (0.59) | 2.33 (0.58)
    AM nasal congestion | 2.57 (0.41) | 2.56 (0.46) | 2.55 (0.45) | 2.56 (0.44)
    PM sneezing | 2.06 (0.68) | 2.10 (0.75) | 2.10 (0.69) | 2.09 (0.71)
    PM runny nose | 2.40 (0.59) | 2.34 (0.63) | 2.35 (0.59) | 2.36 (0.60)
    PM nasal itching | 2.27 (0.62) | 2.30 (0.60) | 2.27 (0.60) | 2.28 (0.60)
    PM nasal congestion | 2.47 (0.49) | 2.47 (0.52) | 2.48 (0.50) | 2.48 (0.50)
    AM and PM sneezing | 2.05 (0.66) | 2.10 (0.72) | 2.08 (0.67) | 2.08 (0.68)
    AM and PM runny nose | 2.41 (0.54) | 2.38 (0.57) | 2.39 (0.55) | 2.39 (0.55)
    AM and PM nasal itching | 2.28 (0.59) | 2.34 (0.55) | 2.29 (0.57) | 2.30 (0.57)
    AM and PM nasal congestion | 2.52 (0.43) | 2.52 (0.47) | 2.52 (0.45) | 2.52 (0.45)
Baseline Instantaneous Nasal Symptom Score (iNSS) [Mean (Standard Deviation); unit: unit on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  unit on a scale
    AM sneezing | 1.73 (0.84) | 1.75 (0.91) | 1.73 (0.88) | 1.74 (0.88)
    AM runny nose | 2.32 (0.58) | 2.26 (0.64) | 2.29 (0.64) | 2.29 (0.62)
    AM nasal itching | 2.22 (0.66) | 2.23 (0.64) | 2.20 (0.68) | 2.22 (0.66)
    AM nasal congestion | 2.50 (0.47) | 2.48 (0.51) | 2.47 (0.53) | 2.48 (0.50)
    PM sneezing | 1.79 (0.82) | 1.79 (0.89) | 1.77 (0.88) | 1.78 (0.86)
    PM runny nose | 2.22 (0.65) | 2.18 (0.69) | 2.16 (0.70) | 2.19 (0.68)
    PM nasal itching | 2.13 (0.68) | 2.17 (0.66) | 2.10 (0.69) | 2.13 (0.67)
    PM nasal congestion | 2.36 (0.54) | 2.36 (0.57) | 2.34 (0.55) | 2.35 (0.55)
    AM and PM sneezing | 1.76 (0.81) | 1.77 (0.86) | 1.75 (0.86) | 1.76 (0.84)
    AM and PM runny nose | 2.27 (0.60) | 2.22 (0.62) | 2.23 (0.64) | 2.24 (0.62)
    AM and PM nasal itching | 2.18 (0.65) | 2.20 (0.61) | 2.15 (0.66) | 2.17 (0.64)
    AM and PM nasal congestion | 2.43 (0.48) | 2.42 (0.51) | 2.41 (0.51) | 2.42 (0.50)
Baseline Individual Reflective Ocular Symptom Score (rOSS) in Subjects with (rTOSS) ≥5.0 [Mean (Standard Deviation); unit: unit on a scale] — OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms.)Reflective OSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  unit on a scale
    AM itching eyes | 2.49 (0.44) | 2.52 (0.43) | 2.48 (0.44) | 2.49 (0.43)
    AM redness of eyes | 2.31 (0.57) | 2.28 (0.62) | 2.24 (0.60) | 2.28 (0.60)
    AM tearing eyes | 2.30 (0.48) | 2.37 (0.51) | 2.28 (0.50) | 2.31 (0.50)
    PM itching eyes | 2.47 (0.45) | 2.50 (0.47) | 2.45 (0.48) | 2.47 (0.47)
    PM redness of eyes | 2.28 (0.58) | 2.26 (0.65) | 2.24 (0.62) | 2.26 (0.62)
    PM tearing eyes | 2.25 (0.56) | 2.34 (0.52) | 2.25 (0.51) | 2.28 (0.53)
    AM and PM itching eyes | 2.48 (0.43) | 2.51 (0.43) | 2.46 (0.44) | 2.48 (0.43)
    AM and PM redness of eyes | 2.29 (0.55) | 2.27 (0.62) | 2.24 (0.59) | 2.27 (0.59)
    AM and PM tearing eyes | 2.27 (0.49) | 2.35 (0.49) | 2.27 (0.48) | 2.30 (0.49)
Baseline Individual Instantaneous Ocular Symptom Score (iOSS) in subjects with (iTOSS) ≥5.0 [Mean (Standard Deviation); unit: unit on a scale] — OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous OSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  unit on a scale
    AM itching eyes | 2.47 (0.43) | 2.47 (0.44) | 2.45 (0.47) | 2.46 (0.44)
    AM redness of eyes | 2.34 (0.56) | 2.29 (0.60) | 2.31 (0.52) | 2.31 (0.56)
    AM tearing eyes | 2.26 (0.50) | 2.32 (0.52) | 2.29 (0.45) | 2.29 (0.49)
    PM itching eyes | 2.41 (0.46) | 2.40 (0.50) | 2.41 (0.47) | 2.41 (0.47)
    PM redness of eyes | 2.30 (0.58) | 2.24 (0.62) | 2.28 (0.54) | 2.27 (0.58)
    PM tearing eyes | 2.19 (0.57) | 2.25 (0.56) | 2.22 (0.48) | 2.22 (0.54)
    AM and PM itching eyes | 2.44 (0.42) | 2.43 (0.44) | 2.43 (0.44) | 2.43 (0.43)
    AM and PM redness of eyes | 2.32 (0.54) | 2.26 (0.58) | 2.29 (0.50) | 2.29 (0.54)
    AM and PM tearing eyes | 2.23 (0.50) | 2.28 (0.50) | 2.26 (0.42) | 2.26 (0.48)
Baseline Rhinoconjunctivitis Quality of Life Questionnaire [RQLQ(S)] ≥3.0 [Mean (Standard Deviation); unit: units on a scale] — RQLQ(S) in subjects with baseline RQLQ[S] score ≥3.0. RQLQ(S) consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
  units on a scale | 4.30 (0.80) | 4.42 (0.87) | 4.36 (0.78) | 4.36 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Subject-reported AM and PM Reflective TNSS Averaged Over the Two-week Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
Units on a scale | -1.74 (0.15) | -1.75 (0.15) | -0.72 (0.16)
Statistical Analysis 1: Comparison: Ciclesonide HFA Nasal Aerosol 160 μg vs Placebo; The null hypothesis is that there is no difference in primary outcome when compare active to placebo group. The alternative hypothesis is that there is a difference in primary outcome when compare active to placebo group. It was estimated that 200 subjects per group will provide at least 85% power to detect a difference between treatment groups of 0.7 in the change from baseline in rTNSS with a two-sided alpha level of 0.025; Test type: Superiority or Other; p < 0.0001, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.59 to 1.45]
Statistical Analysis 2: Comparison: Ciclesonide HFA Nasal Aerosol 80 μg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [0.61 to 1.46]

2. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Instantaneous TNSS Averaged Over the 2-week Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale | -0.36 (0.04) | -0.36 (0.04) | -0.18 (0.04)
Statistical Analysis 1: Comparison: Ciclesonide HFA Nasal Aerosol 160 μg vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.07 to 0.29]
Statistical Analysis 2: Comparison: Ciclesonide HFA Nasal Aerosol 80 μg vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.08 to 0.29]

3. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Reflective TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TOSS symptom scores assess symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
units on a scale | -1.21 (0.13) | -1.40 (0.13) | -0.88 (0.13)
Statistical Analysis 1: Comparison: Ciclesonide HFA Nasal Aerosol 160 μg vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.1444, ANCOVA — Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.03 to 0.71]
Statistical Analysis 2: Comparison: Ciclesonide HFA Nasal Aerosol 80 μg vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.0124, ANCOVA — Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.15 to 0.89]

4. Secondary Outcome: Change From Baseline in the RQLQ(S) Overall Score at the End of the 2-week Treatment Period in Impaired Subjects With Baseline RQLQ(S) Score of ≥3.0
Description: RQLQ(S) in impaired subjects with baseline RQLQ[S] score ≥3.0. RQLQ(S) consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 148 | 162 | 145
units on a scale | -1.41 (0.12) | -1.44 (0.11) | -0.79 (0.12)
Statistical Analysis 1: Comparison: Ciclesonide HFA Nasal Aerosol 160 μg vs Placebo; Test type: Superiority or Other; p = 0.0124, ANCOVA — Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [0.30 to 0.94]
Statistical Analysis 2: Comparison: Ciclesonide HFA Nasal Aerosol 80 μg vs Placebo; Test type: Superiority or Other; ANCOVA — Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [0.33 to 0.95]

5. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Reflective TNSS Averaged Over the 2-week Treatment Period.
Description: as for outcome 1
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale | -1.77 (0.15) | -1.84 (0.15) | -0.77 (0.16)

6. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Reflective TNSS Averaged Over the 2 Week Treatment Period.
Description: as for outcome 1
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale | -1.70 (0.16) | -1.67 (0.16) | -0.66 (0.16)

7. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Instantaneous TNSS Averaged Over the 2-week Treatment Period.
Description: as for outcome 2
Time Frame: Week0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale | -1.56 (0.15) | -1.60 (0.15) | -0.71 (0.15)

8. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Instantaneous TNSS Averaged Over the 2-week Treatment Period.
Description: as for outcome 2
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale | -1.46 (0.16) | -1.56 (0.15) | -0.64 (0.16)

9. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Reflective TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0
Description: as for outcome 3
Time Frame: Week 0-2
Population: In subjects with baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
units on a scale | -1.24 (0.14) | -1.41 (0.14) | -0.88 (0.13)

10. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Reflective TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0
Description: as for outcome 3
Time Frame: Week 0-2
Population: In subjects with baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
units on a scale | -1.21 (0.14) | -1.39 (0.14) | -0.88 (0.14)

11. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Instantaneous TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0.
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In subjects with baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale | -1.12 (0.14) | -1.24 (0.14) | -0.72 (0.14)

12. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Instantaneous TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0.
Description: as for outcome 11
Time Frame: Week 0-2
Population: In subjects with baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale | -1.14 (0.15) | -1.20 (0.15) | -0.74 (0.15)

13. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Instantaneous TOSS Averaged Over the 2-week Treatment Period in Subjects With Baseline TOSS ≥5.0.
Description: as for outcome 11
Time Frame: Week 0-2
Population: In subjects with baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale | -1.13 (0.14) | -1.21 (0.14) | -0.72 (0.14)

14. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Instantaneous NSS Averaged Over the 2-week Treatment Period
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  Sneezing | -0.36 (0.04) | -0.40 (0.04) | -0.14 (0.04)
  Runny Nose | -0.40 (0.04) | -0.45 (0.04) | -0.18 (0.04)
  Nasal Itching | -0.45 (0.04) | -0.39 (0.04) | -0.21 (0.04)
  Nasal Congestion | -0.35 (0.04) | -0.37 (0.04) | -0.18 (0.04)

15. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Instantaneous NSS Averaged Over the 2-week Treatment Period
Description: as for outcome 14
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  Sneezing | -0.35 (0.04) | -0.40 (0.04) | -0.14 (0.04)
  Runny Nose | -0.36 (0.04) | -0.42 (0.04) | -0.16 (0.04)
  Nasal Itching | -0.39 (0.04) | -0.37 (0.04) | -0.16 (0.04)
  Nasal Congestion | -0.36 (0.04) | -0.36 (0.04) | -0.18 (0.04)

16. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Instantaneous NSS Averaged Over the 2-week Treatment Period
Description: as for outcome 14
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  Sneezing | -0.35 (0.04) | -0.40 (0.04) | -0.14 (0.04)
  Runny Nose | -0.38 (0.04) | -0.43 (0.04) | -0.17 (0.04)
  Nasal Itching | -0.42 (0.04) | -0.38 (0.04) | -0.19 (0.04)
  Nasal Congestion | -0.36 (0.04) | -0.36 (0.04) | -0.18 (0.04)

17. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Reflective Nasal Symptom Scores (NSS) Averaged Over the 2-week Treatment Period.
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  sneezing | -0.47 (0.04) | -0.51 (0.04) | -0.18 (0.05)
  runny nose | -0.44 (0.04) | -0.51 (0.04) | -0.21 (0.04)
  nasal itching | -0.47 (0.04) | -0.43 (0.04) | -0.20 (0.04)
  nasal congestion | -0.40 (0.04) | -0.38 (0.04) | -0.18 (0.04)

18. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Reflective NSS Averaged Over the 2-week Treatment Period.
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  Sneezing | -0.43 (0.04) | -0.43 (0.04) | -0.14 (0.04)
  Runny Nose | -0.43 (0.04) | -0.45 (0.04) | -0.16 (0.05)
  Nasal Itching | -0.45 (0.04) | -0.39 (0.04) | -0.16 (0.04)
  Nasal Congestion | -0.39 (0.04) | -0.40 (0.04) | -0.20 (0.04)

19. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Reflective NSS Averaged Over the 2-week Treatment Period.
Description: as for outcome 18
Time Frame: Week 0-2
Population: Intent to Treat Population. Not all subjects analyzed due to missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 225 | 226 | 218
units on a scale
  Sneezing | -0.45 (0.04) | -0.47 (0.04) | -0.16 (0.04)
  Runny Nose | -0.44 (0.04) | -0.41 (0.04) | -0.18 (0.04)
  Nasal Itching | -0.44 (0.04) | -0.41 (0.04) | -0.18 (0.04)
  Nasal Congestion | -0.39 (0.04) | -0.39 (0.04) | -0.19 (0.04)

20. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Instantaneous OSS in Subjects With Baseline TOSS≥5.0
Description: OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Instantaneous OSS measures these symptoms over the previous 10 minute time interval. iTOSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale
  itching eyes | -0.37 (0.05) | -0.39 (0.05) | -0.24 (0.05)
  redness of eyes | -0.38 (0.05) | -0.38 (0.05) | -0.21 (0.05)
  tearing eyes | -0.37 (0.05) | -0.47 (0.05) | -0.27 (0.05)

21. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Instantaneous OSS in Subjects With Baseline TOSS≥5.0
Description: as for outcome 20
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale
  itching eyes | -0.38 (0.05) | -0.37 (0.05) | -0.25 (0.05)
  redness of eyes | -0.39 (0.05) | -0.37 (0.05) | -0.27 (0.05)
  tearing eyes | -0.38 (0.05) | -0.45 (0.05) | -0.22 (0.06)

22. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Instantaneous OSS in Subjects With Baseline TOSS≥5.0
Description: as for outcome 20
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 146 | 141 | 137
units on a scale
  itching eyes | -0.37 (0.05) | -0.38 (0.05) | -0.24 (0.05)
  redness of eyes | -0.39 (0.05) | -0.38 (0.05) | -0.24 (0.05)
  tearing eyes | -0.37 (0.05) | -0.46 (0.05) | -0.24 (0.05)

23. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Reflective OSS in Subjects With Baseline TOSS ≥5.0
Description: OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective OSS measures these symptoms over the previous 12-hour time interval. rTOSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: participants
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
participants
  itching eyes | -0.41 (0.05) | -0.45 (0.05) | -0.31 (0.05)
  redness of eyes | -0.41 (0.05) | -0.42 (0.05) | -0.25 (0.05)
  tearing eyes | -0.42 (0.05) | -0.53 (0.05) | -0.33 (0.05)

24. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Reflective OSS in Subjects With Baseline TOSS ≥5.0
Description: as for outcome 23
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: participants
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
participants
  itching eyes | -0.42 (0.05) | -0.43 (0.05) | -0.28 (0.05)
  redness of eyes | -0.39 (0.05) | -0.42 (0.05) | -0.28 (0.05)
  tearing eyes | -0.40 (0.05) | -0.54 (0.05) | -0.32 (0.05)

25. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Reflective OSS in Subjects With Baseline TOSS ≥5.0
Description: as for outcome 23
Time Frame: Week 0-2
Population: In Subjects With Baseline TOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 161 | 159 | 164
units on a scale
  itching eyes | -0.42 (0.05) | -0.44 (0.05) | -0.29 (0.05)
  redness of eyes | -0.39 (0.05) | -0.42 (0.05) | -0.27 (0.05)
  tearing eyes | -0.41 (0.05) | -0.53 (0.05) | -0.32 (0.05)

26. Secondary Outcome: Change From Baseline in the RQLQ(S) Domains at the End of the 2-week Treatment Period in Impaired Subjects With Baseline RQLQ(S) Score of ≥3.0
Description: RQLQ(S) in subjects with baseline RQLQ[S] score ≥3.0. RQLQ(S) consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
Time Frame: Week 0-2
Population: In Impaired Subjects with Baseline RQLQ(S) Score of ≥3.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Number analyzed (Participants) | 148 | 162 | 145
units on a scale
  Overall Score | -1.41 (0.12) | -1.44 (0.11) | -0.79 (0.12)
  Domain 1: Activities | -1.39 (0.13) | -1.34 (0.12) | -0.70 (0.13)
  Domain 2: Sleep | -1.49 (0.14) | -1.60 (0.13) | -0.83 (0.14)
  Domain 3: Non-Nose/Eye Symptoms | -1.33 (0.12) | -1.21 (0.11) | -0.67 (0.12)
  Domain 4: Practical Problems | -1.62 (0.13) | -1.64 (0.12) | -0.91 (0.13)
  Domain 5: Nasal Symptoms | -1.52 (0.13) | -1.61 (0.12) | -0.83 (0.13)
  Domain 6: Eye Symptoms | -1.25 (0.13) | -1.25 (0.12) | -0.81 (0.13)
  Domain 7: Emotional | -1.36 (0.13) | -1.36 (0.12) | -0.82 (0.13)

27. Secondary Outcome: Time to Maximal Effect Over the 2-week of Double-blind Treatment Period.
Description: The time to maximal effect is defined as the number of days until the first treatment day on which the estimated difference between Ciclesonide HFA and placebo is at least 90% of the largest estimated difference. This is based on the analyses of change from baseline in the average of AM and PM reflective TNSS scores for each day. The evaluation is made separately for each dose level of Ciclesonide HFA compared to placebo.
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg
Number analyzed (Participants) | 225 | 226
Days | 7 (0.18) | 8 (0.19)

ADVERSE EVENTS:
Arm/Group | Ciclesonide HFA Nasal Aerosol 160 μg | Ciclesonide HFA Nasal Aerosol 80 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/226 | 0/220
Other Adverse Events (participants affected / at risk) | 6/225 | 3/226 | 4/220
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide HFA Nasal Aerosol 160 μg (N=225) | Ciclesonide HFA Nasal Aerosol 80 μg (N=226) | Placebo (N=220)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
This study was not designed or powered for a comparison of the 80mcg dose with the 160mcg dose therefore no statistical comparisons were planned between the two active groups. Publication references to 74 and 148mcg are equivalent to 80 and 160mcg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other